CLINICAL TRIAL: NCT05607719
Title: The Effect of Inhaled Corticosteroids (ICS) Adjunct Therapy on Pulmonary Vascular Endothelial Function in Chronic Obstructive Pulmonary Disease (COPD): Comparison of Two Standard Treatments (NCT05607719
Brief Title: Inhaled Corticosteroids (ICS) on Pulmonary Endothelial Function in COPD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Adam Wanner, Professor of Medicine, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 20220347
Record Dates: First submitted 2022-11-02; First posted 2022-11-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bretzri followed by Bevespi Group (Experimental): Participants in this group will receive Bretzri for 4-weeks followed by 8-weeks of Bevespi.
  Interventions: Drug: Bevespi; Drug: Bretzri
- Bevespi followed by Bretzri Group (Experimental): Participants in this group will receive Bevespi for 8-weeks followed by 4-weeks of Bretzri.
  Interventions: Drug: Bevespi; Drug: Bretzri

INTERVENTIONS:
Drug: Bevespi — Two puffs twice a day
Drug: Bretzri — Two puffs twice a day

SUMMARY:
The study objective is to determine whether an ICS added for 4 weeks to a baseline treatment with a Long-Acting Beta-adrenergic Agonist (LABA) and Long-Acting Muscarinic Antagonist (LAMA) combination improves pulmonary vascular endothelial function as assessed by the vasodilator response to inhaled albuterol (endothelium-dependent vasodilation) in stable COPD patients treated with a LABA/LAMA without an ICS for at least one month.

ELIGIBILITY:
Inclusion Criteria:

* physician diagnosis of COPD
* former smoking history of more than 10 pack-years
* baseline post-bronchodilator one-second forced expiratory volume (FEV1) 50-80% of predicted, baseline FEV1 and forced vital capacity (FVC) ratio <0.7
* males and females, 40-80 years of age
* regular use of a LAMA/LABA drug regimen for at least a month

Exclusion Criteria:

* women of childbearing potential who do not use accepted birth- control measures
* pregnant and breast-feeding women
* respiratory infection within 4 weeks of a test day
* a Corona Virus Disease (COVID) vaccination <3 months prior to study entry
* ICS use (within 4 weeks of study entry)
* ICS hypersensitivity
* albuterol intolerance
* use of beta-blocker medication (oral and ophthalmic)
* use of systemic glucocorticosteroid medication within 6 wk prior to the screening visit
* an acute COPD exacerbation within 6 wk of the screening day (defined as a need for antibiotic or systemic glucocorticoid therapy or emergency department (ED) visit/hospitalization)
* current smoking or vaping tobacco or other products
* Oxygen (O2) saturation of <90% at-rest breathing room air
* Long-term oxygen therapy (LTOT) required at rest
* regular use of pulmonary vasodilators
* systemic arterial systolic pressure >150 mmHg and diastolic pressure >100 mmHg on the test day
* a >40mmHg right ventricular systolic pressure (RVSP) by prior echocardiography
* a documented COVID infection within 4 weeks of the screening day
* Regular use of home oxygen at rest
* Physician diagnosis of obesity hypoventilation syndrome

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Albuterol induced percent change in pulmonary vascular resistance (PVR) | baseline to 15 minutes post inhalation
  Echocardiographic assessment of PVR before and after inhalation of 180 μg albuterol as a test of endothelial function

SECONDARY OUTCOMES:
Albuterol induced absolute change in PVR | baseline, up to 45 minutes post inhalation
  Echocardiographic assessment of PVR before and after inhalation of 180 μg albuterol as a test of endothelial function
Percent change in FEV1 | baseline to 15 minutes post inhalation
  Percent change in FEV1 will be measured using spirometry
Change in oxygen saturation | baseline, up to 45 minutes post inhalation
  Change in oxygen saturation measured by pulse oximetry

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wanner, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States